CLINICAL TRIAL: NCT01639716
Title: Aggressive Non-Lymphoma and T Helper 2 Cytokines Relationship With Prognostic Markers
Brief Title: Lymphoma and T Helper 2 Cytokines Relationship With Prognostic Markers
Status: Completed | Type: Observational
Sponsor: Nil Guler (Individual)
Responsible Party: Sponsor-Investigator, Nil Guler, Medical Doctor, Guler, Nil, M.D.
Organization: Guler, Nil, M.D. (Individual)
Other Study IDs: NG63900; NG6420 (Other Grant/Funding Number: NG6420); NG6420 (Other Grant/Funding Number: Nil Guler)
Record Dates: First submitted 2012-07-04; First posted 2012-07-13 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Lymphoma
Keywords: Survey, interleukin status
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Biospecimen Retention: Samples Without DNA — periperal blood sample
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (7):
- Lymphoma group
- healthy group
- IL-10 high
- IL-10 low
- IL-4 high
- IL-4 low
- lymphopenia

SUMMARY:
The investigators hypothesized that Non Hodgkin lymphoma is using T helper 2 pathways. So that the investigators decided to study of cytokines related to T helper 2 pathways. It is well known that parasites and allergic situations also use T helper 2 pathways. Because that the investigators excluded the patients have parasites and allergic situations. All the patients were over 18. The investigators included the patients with non Hodgkin lymphoma which new diagnosed. It is observational study. The investigators took blood before chemotherapy and four months later. The investigators did not interfere with which chemotherapy will be given to patients. This decision was belong to hematologist or oncologist who will treat the patient.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed non hodgkin lymphoma
* Diffuse large B cell lymphoma and T cell lymphoma patients

Exclusion Criteria:

* under 18 age
* parasitosis
* allergic status

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 31 newly diagnosed non hodgkin lymphoma and 27 healthy controls. We studied IL-10 and IL-4 in lymphoma group and healthy group and observed patients till end of study. We analised survival. We compared with IL-4 and IL-10 levels with prognostic factors.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2011-05; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Interleukin 4 and Interleukin 10 levels as pg/mL in non hodgkin lymphoma | This study ended within 13 months
  We will measure 31 patients and 27 healthy person's Interleukin 4 and Interleukin 10 levels as pg/mL at the beginning of the study. We determined all of the patients IPI score, LDH (U/L), crp (mg/L), erythrocyte sedimentation rate, hemoglobin (gr/dL), lymphocyte count in per µL, albumin (gr/dL) before the treatment. We wanted to check whether there is any correlation between well known prognostic markers (LDH, crp, albumin, stage, ECOG performance status) and Interleukin-4 and interleukin-10 levels.

SECONDARY OUTCOMES:
survey as months | During study which was 13 months
  Our secondary goal was to determine the survey time as month from diagnoses to die from any reason or last evaluation during our study which was 13 months.

CONTACTS AND LOCATIONS:
Overall Officials: Nil Guler, MD, Principal Investigator; Nil Guler, MD, Principal Investigator — ONDOKUZ MAYİS UNİVERSİTY, SCHOOL OF MEDİCİNE
Locations (1):
- Ondokuz Mayis University Medical School, Samsun, Atakum, Turkey (Türkiye)

REFERENCES:
- See also: OMU School of Medicine. Contact via e-mail. — http://www.omu.edu.tr